CLINICAL TRIAL: NCT03418818
Title: A Prospective Study of Hypoxia Imaging in Patients With Soft Tissue Sarcoma Using Positron Emission Tomography (PET) With 18F-Fluoroazomycin Arabinoside (18F-FAZA) in Combination With MRI
Brief Title: FAZA PET/MRI Sarcoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-6178
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Sarcoma
Keywords: hypoxia; sarcoma; FAZA; PET Imaging
MeSH Terms: conditions — Sarcoma; Hypoxia | interventions — fluoroazomycin arabinoside; pimonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants will complete FAZA PET/MRI scan and radiation therapy before surgery.
  Interventions: Drug: 18F-FAZA
- Arm B (Experimental): Participants will receive pimonidazole prior to surgery. Participants in Arm B also have the option to complete a FAZA PET/MRI scan prior to surgery.
  Interventions: Drug: Pimonidazole

INTERVENTIONS:
Drug: 18F-FAZA — 18F-FAZA is a radiotracer used for PET imaging (in combination with MRI) to detect hypoxia in tumours. This scan will be done before and after their radiation treatment.
  Arms: Arm A
Drug: Pimonidazole — Pimonidazole is a drug that will attached to areas in the tumour that are low in oxygen. When this occurs, the areas of the tumour that are low in oxygen can be more easily found and studied after surgical removal.
  Arms: Arm B

SUMMARY:
This is a dual arm, single centre, investigator initiated study to investigate the use of FAZA-PET in combination with MRI. FAZA is an investigational radiotracer used in PET scans. FAZA PET/MRI will be used to measure hypoxia in sarcoma tissues and will occur for:

Arm A: before neo-adjuvant radiation/chemotherapy treatment; Arm B: before surgery (optional).

After the FAZA PET/MRI scan, patients will be followed up via telephone, 48 hours after the scan, to see if there are any side effects due to FAZA.

Up to 30 patients enrolled in Arm B will receive pimonidazole approximately 16-20 hours before surgery.

DETAILED DESCRIPTION:
Mutliple studies show that hypoxia in sarcoma has been consistently associated with poor treatment outcomes. Subsequently, there has been a study that shows inhibition of hypoxia-induced transcription factor (HIF-1 alpha), with radiation, was effective in disease treatment in pre-clinical models. This shows how important hypoxia was in playing a role in overall disease outcome and survival.

As a means of examining tumor features, such as hypoxia, hybrid PET/MR imaging combines the advantages of MRI's soft-tissue and contrast resolution with PET's functional metabolic capabilities. There have been few reports of using 18F-FDG in diagnostic PET/MRI. with the use of 18F-FAZA in this study, parameters such as diffusion, micro-perfusion, and contrast enhancement (as a surrogate marker for viable tumour tissue) can be simultaneously compared with the FAZA-derived pattern, in a single procedure.

The study is being conducted to measure the volume of hypoxic tumor in high-risk STS patients, using FAZA-PET/MRI, before and after neoadjuvant radiotherapy/chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with either: high-risk extremity STS (g2-3, > 10 cm largest dimension, and leiomyosarcoma, synovial sarcoma, malignant peripheral nerve sheath tumour, or undifferentiated pleomorphic sarcoma), or: high-risk RPS (g2-3, and leiomyosarcoma or dedifferentiated liposarcoma)
3. Intention to treat using radiotherapy/chemotherapy/surgery according to the current treatment policies of the Sarcoma Site Group of PM
4. A negative serum pregnancy test within the two-week interval immediately prior to PET-MR imaging, for women of child-bearing age
5. Ability to provide written informed consent to participate in the study

Exclusion Criteria:

1. Previous radiotherapy to intended treatment volumes.
2. Previous systemic therapy
3. Active malignancy other than sarcoma
4. Unable to remain supine for at least 60 minutes
5. Pregnancy or breast feeding
6. Age less than 18 years old
7. Failure to provide written informed consent
8. Contraindication for MR as per current institutional guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Grade of FAZA uptake in the primary tumor | 2 years
  Graded based on images from the 2-hour static scan: 0, uptake less than surrounding normal background tissues; 1, no regions of focal uptake higher than that of background; 2, focal uptake moderately higher than background; and 3, focal uptake markedly higher than background

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada